CLINICAL TRIAL: NCT01114321
Title: Glucose Tolerance in Patients With an Idiopathic Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Patrick LACARIN, CHU Clermont-Ferrand
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-0070
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Parkinson's Disease
Keywords: Idiopathic Parkinson's disease; Glucose intolerance; Diabetes; OGTT; Patient with an Idiopathic Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Glucose Intolerance; Diabetes Mellitus | interventions — Proteins; Caloric Restriction

INTERVENTIONS:
Behavioral: Protein and calorie controlled diet — Protein and calorie controlled diet Self-hypnotic relaxation

SUMMARY:
Dysfunction of autonomic nervous system is an important non motor feature of Parkinson' disease (PD). Lewy body formation is widely distributed in hypothalamus and in sympathetic and parasympathetic systems. Animal studies suggest a link between hypothalamus sensing of substrates and glucose metabolism. Thus, hypothalamus lesions could lead to change in glucose metabolism. Recently, we showed that fasting blood glucose level was significantly higher in PD patients than in control group suggesting that glucose tolerance may be impaired in PD. Some studies provided evidence for higher diabetes prevalence in PD patients whereas others showed no difference or a reduced risk of diabetes prevalence in PD patients compared to healthy subjects.

So, the risk that a PD patient develops a glucose intolerance or a diabetes is not clearly established and merit to be studied considering the damageable consequences for patient healthy.

The aim of this prospective study was to determine the risk that a PD patient develop a glucose intolerance or a diabetes compared to a matched control group, using an oral glucose tolerance test (OGTT).

DETAILED DESCRIPTION:
50 patients

Inclusion visit :

* Clinical examination/ Interview on health and medical history
* Complete UPDRS, MMS
* Biologic check up

Protocol :

All patients were studied in the postabsorptive state after a 10-h overnight fast.

On the day of the experiment, patients did not receive their treatment. One catheter was inserted for blood sample collections. Patients ingested then 75 g of glucose.

Blood samples were collected for plasma glucose and plasma insulin concentration analyses at T0, T30, T60, T90, T120, T150 and T180. Urinary glucose was researched at T0 and T120.

In parallel, a dysautonomia evaluation of each patient was made (SCOPA AUT questionnaire, Tilt test).

ELIGIBILITY:
Inclusion Criteria:

* Age : 18-70 years
* Patient with an idiopathic Parkinson's disease according to the criteria of the "Parkinson's Disease Society Brain Bank" with a duration of disease >5years
* MMS>24/30
* No treatment modification 7 days before the inclusion
* Affiliation to social security
* Agreement of patients

Exclusion Criteria:

* Patient treated with antibiotics, AINS, AIS or other treatment which could interfere with the protocol
* Patients with significant heart, respiratory, psychiatric, metabolic, hepatic, kidney diseases; diabetes, heart deficiency, chronic kidney deficiency, untreated thyroid disease …
* Patient treated with a deep brain stimulation
* Patients with metabolic and/or biological anomalies
* Pregnant women
* Medical or chirurgical previous history which could interfere with the protocol
* Alcohol (>30g/day); Tobacco (>10 cigarettes/day)
* Participation to an other study at the same time

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the plasma glucose concentration measured 120 min after the oral glucose surcharge intake. | 120 min after the oral glucose surcharge intake.

SECONDARY OUTCOMES:
Plasma insulin concentration kinetic | at T0, T30, T60, T90, T120, T150 and T180
Plasma glucose concentration kinetic | at T0, T30, T60, T90, T120, T150 and T180
Urinary glucose measurement | at T0 and T120

CONTACTS AND LOCATIONS:
Overall Officials: Franck DURIF, PUPH, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Chu Clermont-Ferrand, Clermont-Ferrand

REFERENCES:
- [Derived] Beze S, Castellani L, Pereira B, Chiambaretta F, Durif F, Marques A. Two-year longitudinal follow-up of visual illusions and hallucinations in Parkinson's disease. J Neurol. 2022 Aug;269(8):4546-4554. doi: 10.1007/s00415-022-11074-2. Epub 2022 Mar 16. PMID 35296961
- [Derived] Marques A, Beze S, Pereira B, Chassain C, Monneyron N, Delaby L, Lambert C, Fontaine M, Derost P, Debilly B, Rieu I, Lewis SJG, Chiambaretta F, Durif F. Visual hallucinations and illusions in Parkinson's disease: the role of ocular pathology. J Neurol. 2020 Oct;267(10):2829-2841. doi: 10.1007/s00415-020-09925-x. Epub 2020 May 23. PMID 32447550
- [Derived] Marques A, Dutheil F, Durand E, Rieu I, Mulliez A, Fantini ML, Boirie Y, Durif F. Glucose dysregulation in Parkinson's disease: Too much glucose or not enough insulin? Parkinsonism Relat Disord. 2018 Oct;55:122-127. doi: 10.1016/j.parkreldis.2018.05.026. Epub 2018 May 31. PMID 29866628